CLINICAL TRIAL: NCT00028496
Title: Phase I Study of a Recombinant Fowl Pox Vaccine rF-CEA (6D)/TRICOM Alone or With GM-CSF in Patients With Advanced CEA Expressing Adenocarinomas
Brief Title: Vaccine Therapy With or Without Sargramostim in Treating Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02433; FCCC-01016; CDR0000069093 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Gallbladder; Adenocarcinoma of the Pancreas; Adenocarcinoma of the Rectum; Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Cholangiocarcinoma of the Gallbladder; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Male Breast Cancer; Mixed Adenocarcinoma of the Stomach; Ovarian Endometrioid Adenocarcinoma; Paget Disease of the Breast With Intraductal Carcinoma; Paget Disease of the Breast With Invasive Ductal Carcinoma; Recurrent Adult Primary Liver Cancer; Recurrent Breast Cancer; Recurrent Colon Cancer; Recurrent Gallbladder Cancer; Recurrent Gastric Cancer; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Pancreatic Cancer; Recurrent Rectal Cancer; Recurrent Salivary Gland Cancer; Salivary Gland Adenocarcinoma; Stage II Malignant Testicular Germ Cell Tumor; Stage II Pancreatic Cancer; Stage III Colon Cancer; Stage III Gastric Cancer; Stage III Malignant Testicular Germ Cell Tumor; Stage III Pancreatic Cancer; Stage III Rectal Cancer; Stage III Salivary Gland Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Gastric Cancer; Stage IV Pancreatic Cancer; Stage IV Rectal Cancer; Stage IV Salivary Gland Cancer; Thyroid Gland Medullary Carcinoma; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular; Breast Neoplasms, Male; Breast Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Testicular Neoplasms; Pancreatic Neoplasms; Salivary Gland Neoplasms; Carcinoma, Medullary | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (1):
- Treatment (vaccine therapy, sargramostim, vaccine adjuvant) (Experimental): The first three cohorts of 3-12 patients receive escalating doses of recombinant fowlpox-CEA-TRICOM vaccine (fCEA-TRI) until the maximum tolerated dose (MTD) is determined. fCEA-TRI is administered intradermally every 2 weeks for 4 doses and then every 2 months thereafter (beginning on day 56) in the absence of disease progression or unacceptable toxicity.
  The fourth and fifth cohorts of 6 patients receive fCEA-TRI at the MTD in the same manner as the first three cohorts combined with escalating doses of sargramostim (GM-CSF). GM-CSF is administered subcutaneously once daily beginning on the day of each vaccination and continuing for a total of 4 days.
  The sixth through eighth cohorts of 6 patients receive fCEA-TRI at the MTD in the same manner as the first three cohorts combined with escalating doses of recombinant fowlpox-GM-CSF (rF-GM-CSF).
  Interventions: Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Biological: sargramostim; Biological: recombinant fowlpox GM-CSF vaccine adjuvant

INTERVENTIONS:
Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine — Given intradermally
  Other Names: fowlpox-CEA-B7-1/ICAM-1/LFA-3; rF-CEA(6D)TRICOM
Biological: sargramostim — Given subcutaneously
  Other Names: GM-CSF; Leukine; Prokine
Biological: recombinant fowlpox GM-CSF vaccine adjuvant — Given intradermally
  Other Names: fowlpox-GM-CSF; fowlpox-sargramostim; rf-GM-CSF; rf-sargramostim

SUMMARY:
Phase I trial to study the effectiveness of vaccine therapy with or without sargramostim in treating patients who have advanced or metastatic cancer. Vaccines may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood. Combining vaccine therapy with sargramostim may make tumor cells more sensitive to the vaccine and may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxicity of recombinant fowlpox-CEA-TRICOM vaccine with or without sargramostim (GM-CSF) or recombinant fowlpox-GM-CSF in patients with advanced or metastatic CEA-expressing adenocarcinomas.

II. Determine the CEA-specific T-cell precursor frequency in patients treated with these regimens.

III. Assess the immunogenicity of GM-CSF in patients treated with these regimens.

IV. Determine the inflammatory response and cytokine expression at the vaccination site in these patients 48 hours after vaccination.

V. Correlate telomere length of leukocytes with prior cytotoxic therapies and immunologic response in patients treated with these regimens.

OUTLINE: This is a dose-escalation study. The first three cohorts of 3-12 patients receive escalating doses of recombinant fowlpox-CEA-TRICOM vaccine (fCEA-TRI) until the maximum tolerated dose (MTD) is determined.

The MTD is defined as the dose preceding that at which 2 of 6 patients or 3 of 12 patients experience dose-limiting toxicity. fCEA-TRI is administered intradermally every 2 weeks for 4 doses and then every 2 months thereafter (beginning on day 56) in the absence of disease progression or unacceptable toxicity.

The fourth and fifth cohorts of 6 patients receive fCEA-TRI at the MTD in the same manner as the first three cohorts combined with escalating doses of sargramostim (GM-CSF). GM-CSF is administered subcutaneously once daily beginning on the day of each vaccination and continuing for a total of 4 days.

The sixth through eighth cohorts of 6 patients receive fCEA-TRI at the MTD in the same manner as the first three cohorts combined with escalating doses of recombinant fowlpox-GM-CSF (rF-GM-CSF). rF-GM-CSF is administered in the same manner as GM-CSF.

Patients are followed every month for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma that failed standard curative options and for which no standard palliative options are required within the next 8weeks

  * Advanced or metastatic disease
  * Recurrent or unresectable disease
  * Microscopic metastatic disease confirmed by surgical exploration allowed
* CEA expression by immunohistochemistry
* Circulating CEA greater than 5 ng/mL
* HLA phenotyping required

  * HLA phenotyping must be repeated for patients who have undergone allogeneic bone marrow transplantation
* No clinically symptomatic brain metastases

  * Patients with brain metastases who have completed palliative radiotherapy and have discontinued steroids are eligible
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-1
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST and ALT less than 3 times ULN
* PT and PTT less than 1.5 times ULN (unless therapeutically anticoagulated)
* Creatinine less than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min
* Proteinuria or hematuria less than +2 on urinalysis*
* Urine protein less than 1,000 mg/24-hour collection, if proteinuria greater than +1
* No frequent vomiting or severe anorexia
* No more than 10% weight loss within the past 3 months
* No inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis
* No uncontrolled seizure disorders
* No encephalitis
* No multiple sclerosis
* No allergy to eggs
* No HIV-associated opportunistic infection
* No autoimmune diseases, including the following:

  * Systemic lupus erythematosus
  * Sjögren's syndrome
  * Scleroderma
  * Myasthenia gravis
  * Goodpasture syndrome
  * Addison's disease
  * Hashimoto's thyroiditis
  * Graves' disease
* Antinuclear antibody positive status allowed if no evidence of an autoimmune disease
* No direct contact of vaccination site with the following persons for at least 72 hours after each vaccination:

  * Children under 1 year of age
  * Pregnant women
  * Individuals with eczema or other open skin condition
  * Immunocompromised individuals
* No other concurrent serious medical illness that would preclude study entry
* No other malignancy within the past 2 years except excised basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 1 month before (female patients only), during, and for at least 3 months after study participation
* See Disease Characteristics
* No prior CEA-directed active immunotherapy
* Prior CEA-directed antibody therapy allowed
* At least 4 weeks since prior immunotherapy and recovered
* No other concurrent antineoplastic biologic therapy or immunotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent antineoplastic chemotherapy
* See Disease Characteristics
* No concurrent antineoplastic hormonal therapy
* No concurrent systemic steroids (inhaled steroids allowed)
* Concurrent systemic mineralocorticoids (e.g., megestrol for appetite stimulation or fludrocortisone) allowed
* Concurrent birth control pills allowed
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 50% of all nodal groups
* See Disease Characteristics
* Recovered from prior surgery
* No prior splenectomy
* Concurrent non-steroidal anti-inflammatory drugs allowed
* No other concurrent anti-cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-11; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of recombinant fowlpox-CEA(6D)/TRICOM vaccine determined by dose-limiting toxicities graded according to NCI Common Toxicity Criteria, version 2.0 | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States